CLINICAL TRIAL: NCT03653975
Title: Clinical Features and Potential Etiology of Epilepsy and Nodding Syndrome in the Mahenge Area, Ulanga District
Acronym: NSEC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Thomas Wagner, MD, Heidelberg University
Other Study IDs: HD-DZIF-MUHAS
Record Dates: First submitted 2017-01-25; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Nodding Syndrome; Epilepsy; Onchocerciasis; Cognitive Impairment
Keywords: Nodding Syndrome; Head Nodding; Epilepsy; Onchocerciasis; Cognitive impairment; Mahenge
MeSH Terms: conditions — Nodding Syndrome; Epilepsy; Onchocerciasis; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — To further describe the clinical features of NS, a complete physical and neurological examination in patients with NS and controls is performed at the Mahenge Epilepsy Clinic. All individuals will have to undergo sampling of blood and skin snips from at least two different areas of the body, one of which must be close to the head. Time expenditure for the individual participant is estimated with 60 min (Introduction of the study, consent, skin snip, lumbar puncture and venipuncture) extended for about 60 minutes if EEG recordings are obtained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Nodding syndrome: I) probable Case of Nodding Syndrom (according to the "WHO epidemiologic surveillance case definition") *reported head nodding ** in a previously healthy person with at least 2 major and 1 minor criteria
  Major criteria
  * Age 3 to 18 y at onset of head nodding
  * Nodding frequency 5 to 20 times per min
  Minor criteria
  * Other neurologic abnormalities
  * Clustering in space or time with similar cases
  * Triggering by eating or cold weather
  * Delayed sexual or physical development
  * Psychiatric manifestations
    * As agreed upon at the first International Conference on Nodding Syndrome, Kampala, Uganda, July 2012 (16). ** Repetitive involuntary drops of the head toward the chest on >2 occasions.
  Interventions: Other: no intervention
- epilepsy and onchocerciasis: II) People with epilepsy (PWE) and onchocerciasis (n= 50)
  * confirmed or suspected generalized and idiopathic epilepsy
  * confirmed active infection with O. volvulus (microscopy, PCR and serology)
  Patients with cardiovascular or renal comorbidities, a history of birth or traumatic brain injuries, psychiatric comorbidities, insecure comprehension of the information given, lacking or withdrawn consent will be excluded.
  Interventions: Other: no intervention
- epilepsy, no onchocerciasis: III) People with epilepsy (PWE) without onchocerciasis (n= 50)
  * confirmed or suspected generalized and idiopathic epilepsy
  * excluded active or past infection with O. volvulus (microscopy, PCR and serology)
  Patients with cardiovascular or renal comorbidities, a history of birth or traumatic brain injuries, psychiatric comorbidities, insecure comprehension of the information given, lacking or withdrawn consent will be excluded.
  Interventions: Other: no intervention
- no epilepsy but onchocerciasis: IV) Controls with onchocerciasis, otherwise healthy (n= 50)
  * no evidence for epilepsy or other neurological diseases
  * confirmed active infection with O. volvulus (microscopy, PCR and serology)
  Patients with cardiovascular or renal comorbidities, a history of birth or traumatic brain injuries, psychiatric comorbidities, insecure comprehension of the information given, lacking or withdrawn consent will be excluded.
  Interventions: Other: no intervention
- no epilepsy, no onchocerciasis: V) Healthy Controls without onchocerciasis (n= 50)
  * no evidence for epilepsy or other neurological diseases
  * excluded active or past infection with O. volvulus (microscopy, PCR and serology)
  Patients with cardiovascular or renal comorbidities, a history of birth or traumatic brain injuries, psychiatric comorbidities, insecure comprehension of the information given, lacking or withdrawn consent will be excluded.
  Interventions: Other: no intervention
- controls for Wechsler Nonverbal (WNV): Healthy Controls for cognitive assessment only, (n= 750)
  no evidence for epilepsy or other neurological diseases no detailled examination on O. volvulus performed
  Patients with cardiovascular or renal comorbidities, a history of birth or traumatic brain injuries, psychiatric comorbidities, insecure comprehension of the information given, lacking or withdrawn consent will be excluded.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Background: Childhood epilepsy disorders are particular frequent in the area around Mahenge, southern Tanzania and recent studies have described a novel type of epilepsy with repetitive head nodding episodes and often progressive cognitive dysfunction. Despite the disease affecting thousands in Tanzania, Uganda and South Sudan, etiology and pathogenesis of the disorder termed Nodding Syndrome (NS) is still obscure as the phenotype remains imprecisely described. Epidemiological associations with Onchocerca volvulus and Mansonella spp. were noted at different African sites and remain robust even though no evidence for the presence of O. volvulus in CSF or any previous contact with the CSF was found.

Hypothesis: With regard to the complex host immune reaction to O. volvulus, the investigators hypothesize that the immune response against filariae might contribute to NS and epilepsy. The investigators further assume that specific genetic traits might play a role in the pathogenesis of NS.

Aims In the present study the investigators aim to examine if and how O. volvulus and/or Mansonella spp. contribute to the pathology of NS/epilepsy and therefore intend to analyze the filarial infection and the host immune response in affected children. To identify inherited traits predisposing for epilepsy, NS or specific immune responses, a genetic workup that includes whole-exome sequencing (WES) is performed. The clinical and EEG characteristics are further defined. Cognitive impairment of people with epilepsy and NS is assessed using the Wechsler Nonverbal Scale of Ability (WNV).

Study design: A cross-sectional observational (groups I-III) and a case-control (groups I-V) study recruiting in total 250 patients and controls (I: people with NS, n=50; II: people with epilepsy (PWE) and onchocerciasis, n=50; III: PWE without onchocerciasis, n=50; IV: controls with onchocerciasis but otherwise healthy, n= 50; healthy controls without evidence for onchocerciasis, n= 50) is performed to describe the clinical characteristics in children with NS/epilepsy and to evaluate differences in infection and immune response between groups, respectively. The WNV should be validated in 500 healthy controls to obtain reference data in rural Africa.

Summary: In summary, the study aims to elucidate clinical characteristics and the pathogenesis of NS/epilepsy in children of southern Tanzania and role of parasitic infection as a cause for NS/epilepsy.

DETAILED DESCRIPTION:
Childhood epilepsy disorders are particular frequent in low income countries and especially common in the area around Mahenge, Ulanga region, southern Tanzania, with an epilepsy prevalence of up to 39 per 1000 inhabitants. Therefore, in 1959 Prof. Louise Jilek-Aall founded the Mahenge Epilepsy Clinic to provide basic care to people suffering from convulsive disorders and to enable further in-depth investigations regarding epilepsy. In the summer of 2005, a multinational a team of researchers including the founder of the clinic, Prof. Louise Jilek-Aall, Prof. Erich Schmutzhard, Dr. Andrea Winkler and Prof. William Matuja performed several in-depth etiological investigations. In intensive field research they were able to examine a large number of clinic patients and healthy controls, perform electro-encephalographic and magnetic resonance studies and collect biological materials, such as blood, cerebrospinal fluid (CSF) and skin samples for further sophisticated laboratory tests in Europe. Among others, the studies confirmed the presence of a new type of childhood epilepsy with repetitive head nodding episodes and often progressive cognitive dysfunction. Even though the disease termed Nodding Syndrome (NS) affects thousands in Tanzania, Uganda and South-Sudan, clinical, metabolic and EEG phenotypes are still imprecisely described, and etiology and pathogenesis remain obscure. The high familial occurrence and clustering within circumscribed villages and tribes suggests that genetic traits might play a role. Epidemiological associations with Onchocerca volvulus and Mansonella spp. were noted at different African sites. Despite lacking evidence for the presence of O. volvulus in the CSF the association to NS remains robust.

This is basis for the present study where the investigators aim to examine if and how O. volvulus and/or Mansonella spp. contribute to the pathology of NS, elucidate associated genetic traits, further specify the clinical, metabolic and EEG phenotypes. The investigators will use a cross-sectional observational design including children with NS and epilepsy in order to describe the clinical characteristics and a case-control design to evaluate associated factors.

It is intended to enroll 250 patients and controls between 3 and 18 years of age (I: people with NS, n=50 (inclusion according to the WHO case definition from the first "International Conference on Nodding Syndrome", Kampala, Uganda, July 2012); II: people with epilepsy (PWE) and onchocerciasis, n=50; III: PWE without onchocerciasis, n=50; IV: controls with onchocerciasis but otherwise healthy, n= 50; healthy controls without evidence for onchocerciasis, n= 50). Patients with cardiovascular or renal comorbidities, a history of birth or traumatic brain injuries, lacking or withdrawing consent will be excluded. Groups II to V will be matched to Group I for age, gender and social status.

The investigators intend to analyze the filarial infection and host immune response in affected children compared to unaffected controls. PCR assays will be performed to characterize Onchocerca and Mansonella spp. strains found in patients with NS/PWE and determine Wolbachia loads and features. A novel unique biomarker, N-acetyltyramine-O,ß-glucuronide (NATOG) will be determined to quantify infection with O. volvulus and correlated with other markers that define the host immune response and immune regulation (e.g. regulatory T cells (Treg), cytokines). As polymorphisms in the multidrug-resistance gene 1 (MDR-1) that alter p-glycoprotein expression or function may enhance neurotoxicity of widely used antihelmintic drugs, single nucleotide polymorphism (SNP)-arrays will be determined to investigate if specific polymorphisms might be associated with NS. In addition, the investigators aim to define the clinical picture and course of NS and conduct further EEG investigations and validated neuropsychological tests, follow up patients of previous studies and perform metabolic analyses to specify the metabolic characteristics of NS. A genetic workup that includes whole-exome sequencing (WES) to identify traits predisposing to epilepsy, NS or specific immune responses is scheduled.

In summary, the study aims to elucidate factors that contribute to the high prevalence of NS and epilepsy in the Mahenge area in Southern Tanzania. Also, the research project will have immediate benefits for the population under investigation as people newly diagnosed with epilepsy will be offered treatment at the Mahenge Epilepsy Clinic and staff, patients and relatives will receive further education regarding epilepsy, thereby contributing to sustainability of a standardized approach to care for children with NS and PWE. Conclusions drawn from our study will not only relate to the Mahenge area, but may be applicable to vast numbers of children with NS (northern Uganda and South Sudan) and PWE in other areas. Dissemination of the data through scientific meetings and publications may stimulate further research regarding risk factors for epilepsy in the low income countries.

ELIGIBILITY:
I) Patients with Nodding syndrome confirmed or suspected Case of Nodding syndrome (according to the WHO epidemiologic surveillance case definition: reported head nodding in a previously healthy person with at least 2 major and 1 minor criteria Major criteria Age 3 to 18 y at onset of head nodding Nodding frequency 5 to 20 times per min Minor criteria Other neurologic abnormalities (cognitive decrease, school dropout due to cognitive or behavioral problems, other seizures or neurologic abnormalities) Clustering in space or time with similar cases Triggering by eating or cold weather Delayed sexual or physical development Psychiatric manifestations

As agreed upon at the first International Conference on Nodding Syndrome, Kampala, Uganda, July 2012 (16). EEG,

II) People with epilepsy (PWE) and onchocerciasis confirmed or clinically suspected generalized and idiopathic epilepsy confirmed active infection with O. volvulus (microscopy, PCR and serology)

III) People with epilepsy (PWE) without onchocerciasis confirmed or clinically suspected generalized and idiopathic epilepsy excluded active or past infection with O. volvulus (microscopy, PCR and serology)

IV) Controls with onchocerciasis, otherwise healthy no evidence for epilepsy or other neurological diseases confirmed active infection with O. volvulus (microscopy, PCR and serology)

V) Controls without onchocerciasis, otherwise healthy no evidence for epilepsy or other neurological diseases excluded active or past infection with O. volvulus (microscopy, PCR and serology)

VI) Healthy controls for cognitive assessment, matched to Groups I to V

inclusion criteria: The study groups with their respective inclusion criteria are defined above.

Patients of group I-III will be first recruited into the cross-sectional study and subsequently into the case-control study. Groups II to VI will be matched to Group I for age, gender, social status and stay within the Mahenge area.

exlusion criteria: Patients with evidence for co-infections with HIV, Tb, Malaria or other parasites, cardiovascular or renal comorbidities, a history of birth or traumatic brain injuries, psychiatric comorbidities, insecure comprehension of the information given, lacking or withdrawn consent will be excluded.

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: With support of the hospital staff, participants aged 3 to 99 years will be recruited consecutively among the registered patients as they are seen once a month for a clinical check-up and to receive their medication. Suitable relatives of patients will also be asked to take part in the study.
  The study groups with their respective inclusion criteria are defined above. Patients of group I-III will be first recruited into the cross-sectional study and subsequently into the case-control study. Groups II to VI will be matched to Group I for age, gender, social status and stay within the Mahenge area.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2014-10 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Describing clinical features in children with Nodding Syndrome and other forms of epilepsy e.g. characteristics of the seizures, EEG abnormalities and reporting co-morbidities and impairments. | 2014-2018
  Obtaining clinical features and medical history. Comparing medical history, Seizure types and -frequency and other clinical Features between the groups.
Describing EEG features in children with Nodding Syndrome and other forms | 2014-2018
  Performing EEG recordings and comparing EEG abnormalities (numbers, types and site of epileptiform discharges (ED), background alterations) between the groups.

SECONDARY OUTCOMES:
Measuring the rate of filarial infections in patients with NS, epilepsy and controls. | 2014-2018
  Performing skin snip microscopy and PCR analysis to detect O. volvulus and Mansonella spp. in patients with NS, epilepsy and controls.
Characterization of O. volvulus in patients with Nodding Syndrome and epilepsy. | 2014-2018
Characterization of the host immune response to O. volvulus. | 2014-2018
Analyzing for genetic traits associated with epilepsy, NS, enhanced Ivermectin toxicity or specific immune responses. | 2014-2018
  Performing a genetic workup for known monogenetic forms of epilepsy, single nucleotide polymorphisms (SNP) associated with enhanced Ivermectin toxicity and adverse immune reactions. Performing a Whole-exome sequencing (WES) with biomedical analysis.
Measuring the cognitive impairment in patients with NS and epilepsy. | 2014-2018
  Using the Wechsler Nonverbal Scale of Ability (WNV) and comparing the results to matched healthy controls.

CONTACTS AND LOCATIONS:
Locations (1):
- Mahenge Epilepsy Clinic, Mahenge, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arndts K, Kegele J, Massarani AS, Ritter M, Wagner T, Pfarr K, Lammer C, Dormann P, Peisker H, Menche D, Al-Bahra M, Prazeres da Costa C, Schmutzhard E, Matuja W, Hoerauf A, Layland-Heni LE, Winkler AS. Epilepsy and nodding syndrome in association with an Onchocerca volvulus infection drive distinct immune profile patterns. PLoS Negl Trop Dis. 2023 Aug 3;17(8):e0011503. doi: 10.1371/journal.pntd.0011503. eCollection 2023 Aug. PMID 37535695